CLINICAL TRIAL: NCT02281968
Title: An NSAID Pain Protocol Provides Adequate Pain Relief in Ankle Fractures Treated Operatively
Brief Title: NSAIDs for Pain After Ankle Fracture Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 13-391A
Record Dates: First submitted 2014-10-31; First posted 2014-11-04 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Closed Fracture of Ankle
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NSAID cohort (Experimental): Patients who have had surgical management of ankle fracture will be given a standing regimen (scheduled doses) of 500 mg naproxen twice a day and will have received one intraoperative dose of ketorolac. Patients will have a prescription for opioids for breakthrough pain.
  Interventions: Drug: Naproxen
- Placebo cohort (Placebo Comparator): Patients who have had surgical management of ankle fracture will be given a standing regimen (scheduled doses) of placebo twice a day and will have received one intraoperative dose of saline solution. Patients will have a prescription for opioids for pain.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naproxen — Standing regimen of naproxen in experimental group to reduce need for narcotic to control pain
  Other Names: Naproxen sodium; Naprosyn; Aleve; Anaprox
  Arms: NSAID cohort
Drug: Placebo
  Arms: Placebo cohort

SUMMARY:
The purpose of this study is to investigate if it is possible to decrease opioid consumption in patients undergoing ankle fracture surgery by providing scheduled doses of nonsteroidal inflammatory drugs (NSAIDs). This is a prospective, randomized, double-blinded, placebo controlled study with two groups of patients: one getting NSAIDs to take at regularly scheduled times plus a traditional prescription for opioid medication and one receiving the traditional prescription for opioid medication and a placebo. Patients will be assigned to a group from a computer-generated program. Neither the patients nor their doctors or nurses will know what group they are in, only the pharmacist will have that information. Patients in both groups will have the opportunity to take opioid medications if the pain becomes unmanageable.

DETAILED DESCRIPTION:
Rationale: Opioid abuse is rampant, can have bad consequences, and is a source of many individual and societal problems. Although its use fulfills a role in pain control, this investigation seeks to find a pain control alternative with the potential for fewer adverse consequences for patient undergoing surgery for ankle fracture.

Hypothesis: A structured regimen of NSAIDs (drugs such as ibuprofen or naproxen) during and after ankle fracture surgery will provide adequate pain relief and cause patients to take fewer doses of opioid drugs.

Methods: This will be a prospective, randomized, double-blinded, placebo controlled study of patients with ankle fractures who require surgical treatment by several NSLIJ orthopaedic surgeons at North Shore University Hospital and Long Island Jewish Medical Center. There will be two groups of patients: one getting NSAIDs to take at regularly scheduled times plus a traditional prescription for opioid medication and one receiving the traditional prescription for opioid medication and a placebo. Patients will be assigned to a group from a computer-generated program. Neither the patients nor their doctors or nurses will know what group they are in, only the pharmacist will have that information. Patients in both groups will have the opportunity to take opioid medications if the pain becomes unmanageable. We are evaluating whether patients in the NSAIDs group will a) have no more pain than patients who are prescribed opioid pain killers for the same surgery and b) if the amount of opioid pain killers can be reduced by having patients take scheduled doses of NSAIDs. We will also describe how well or poorly patients heal, looking at several timepoints after surgery, using Xrays to evaluate formation of new bone.

The test (experimental) group will be given a dose of IV (intravenous) ketorolac, which is an NSAID, during surgery, and will be given naproxen 500mg orally two times per day to take on a regular basis after surgery for four weeks. This group will be given percocet 5/325 (an opioid medication) 1-2 pills orally every 4 hours to take as pain medication if the naproxen is not providing adequate pain relief.

The control group will be administered a saline dose during surgery as an equivalent to the IV ketorolac. These patients will take placebo pain pills on a regular basis two times per day for four weeks, and will take percocet for pain relief. This is equivalent to the common pain protocol that is given to patients after ankle fracture surgery, where they are given percocet to be taken on an as-needed basis.

The placebo and naproxen medication will be in unidentifiable capsule form in unmarked bottles. The maximum daily dose of percocet will be 8 pills, so as not to exceed 2.6g acetaminophen daily.

Both groups will take aspirin (ASA) 325mg orally daily for two weeks to prevent blood clots. All patients will take pantoprazole 40mg orally once daily. Pantoprazole is a proton pump inhibitor (PPI) that suppresses the production of stomach acid, to prevent the development of gastrointestinal ulcers.

We will collect demographic data about the patients. We will also collect data about the surgery: surgery time, treating surgeon, type of surgery, location and complexity of fracture.

W are studying the following outcomes: pain relief, opioid use and bone healing. To measure these outcomes, we will use a pain scale called the VAS to look for differences between the group. A change of 10 millimeters on a scale of 100 millimeters will considered to be the important pain difference. We will also ask patients to fill out journals of their medication use, we will perform pill counts, examine Xrays and ask patients to respond to the FFI, a questionnaire to evaluate how well they are functioning.

Patients will be seen for followup at 2 weeks, 6 weeks, 2 months, 6 months, and 1 year after surgery, all but the last visit are the usual and standard visits scheduled after ankle fracture surgery. At each visit, Xrays will be taken of the ankle to evaluate ankle position, and to determine whether bone healing has occurred. Patients will not incur any extra expense as a result of participating in the study.

Since patients will not know which group they have been assigned to -- test (experimental) or control -- the investigators will carefully explain how to determine the need for taking the prescribed opioid pain medication such that patients are not subjected to unnecessary pain. Since both groups will have access to opioid pain medications, the study is designed to determine if those patients in the NSAIDs group already getting the relief from pain will experience pain at lower levels, which we will only be able to determine after the study is completed and the blind is broken.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Sustained an operative ankle fracture that will be treated at Long Island Jewish Medical Center or North Shore University Hospital

Exclusion Criteria:

1. Open fracture
2. Pregnant women
3. Nursing women
4. Dementia
5. Cognitive compromise requiring legal authorized representative Prisoners
6. Uncontrolled hypertension
7. History of peptic ulcer disease
8. Renal insufficiency
9. History of renal transplant
10. eGFR less than 60 mL/min/1.73 m2
11. Chronic liver disease
12. Blood thinners: vitamin K antagonist, factor Xa inhibitors, heparinoids
13. Chronic steroids
14. Immunosuppressive drugs
15. Inflammatory bowel disease
16. Contraindication/allergy for NSAIDs
17. Positive status for HIV
18. Dixogin
19. Methotrexate
20. Vismodebig

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | twelve months
  opioid equivalents
Pain scores | twelve months
  Visual analog scores

SECONDARY OUTCOMES:
bone healing | 12 months
  At each scheduled timepoint from visits 1 through 5, Xrays will be taken of the ankle to evaluate ankle position, and to determine presence and degree of bridging callus on four cortices to evaluate bone healing as a precursor to bony union.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel T. Goldman, MD, Principal Investigator — Northwell Health